CLINICAL TRIAL: NCT00450268
Title: Analysis of Dendritic Cells in Patients Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Dendritic Cells in Patients Following Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: DCalloTX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Other Study IDs: EK208122001
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Last update posted 2007-03-22 (Estimated); Status verified 2007-03

CONDITIONS: Graft Versus Host Disease
Keywords: Graft versus host disease; Allogeneic hematpoietic stem cell transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: blood draw, skin shave biopsy

SUMMARY:
We plan to investigate prospectively and simultaneously skin and blood DC subtypes, their donor/recipient origin and the correlation of DC reconstitution kinetics with treatment, clinical outcome and incidence of aGvHD in patients undergoing allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Blood and skin DC reconstitution shall be investigated in patients affected by hematological diseases and receiving HLA-matched, mobilized peripheral blood stem cells from related or unrelated donors. We plan to simultaneously collect and process double biopsies, i.e. from graft versus host disease affected and non-lesional skin of patients at onset of acute graft versus host disease following allogeneic hematopoietic stem cell transplantation. Emigration assay, Chimerism analysis and immunohistochemistry will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing an allogeneic hematopoietic stem cell transplantation
* Older than 18 years
* WHO-Performance-Status 0 to3
* Informed consent
* Graft versus host disease of the skin

Exclusion Criteria:

* Clotting parameters more than double of normal
* Infection of the skin
* Leucocytes < 1000/µl; Thrombocytes < 20 000/µl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-01; Study Completion 2010-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Gretzinger, MD, Principal Investigator — Universität Carl Gustav Carus Med Klinik I
Locations (1):
- Universitätsklinik Carl Gustav Carus, Dresden, Germany